CLINICAL TRIAL: NCT02925923
Title: The Effects of Crushed Ticagrelor Versus Eptifibatide Bolus +Clopidogrel in Troponin-Negative ACS Patients Undergoing Coronary Intervention
Brief Title: Crushed Ticagrelor Versus Eptifibatide Bolus + Clopidogrel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Massoud Leesar, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F151006002
Record Dates: First submitted 2016-09-27; First posted 2016-10-06 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-02

CONDITIONS: Acute Coronary Syndrome; Angina, Unstable
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable | interventions — Ticagrelor; Eptifibatide; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Active Comparator): crushed ticagrelor (180 mg); (n=50 patients)
  Interventions: Drug: Ticagrelor
- Eptifibatide bolus+clopidogrel (Active Comparator): Eptifibatide bolus (180 mcg/kg x 2 boluses) + clopidogrel 600 mg and heparin low-dose (n=50 patients)
  Interventions: Drug: Eptifibatide; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — After randomization, a blood sample will be obtained at baseline for platelet function study, the study drugs, crushed ticagrelor will be administered. Patients will undergo PCI using drug-eluting stents or bare-metal stents. Blood samples will be obtained at 30 mins, 2, 4, and 24 h after PCI for platelet function tests.
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Eptifibatide — After randomization, a blood sample will be obtained at baseline for platelet function test, the study drugs, clopidogrel and eptifibatide bolus will be administered. Patients will undergo PCI using drug-eluting stents or bare-metal stents. Blood samples will be obtained at 30 mins, 2, 4, and 24 h after PCI for platelet function tests.
  Other Names: Integrilin
  Arms: Eptifibatide bolus+clopidogrel
Drug: Clopidogrel
  Other Names: Plavix
  Arms: Eptifibatide bolus+clopidogrel

SUMMARY:
Patients with troponin-negative acute coronary syndrome (ACS) are not routinely pre-treated with P2Y12 inhibitors and the rate of high on-treatment platelet reactivity (HPR) remains elevated after a loading dose of ticagrelor at the time of percutaneous coronary intervention (PCI). This suggests that faster platelet inhibition with crushed ticagrelor , eptifibatide , or cangrelor is needed to reduce HPR and periprocedural myocardial infarction and injury (PMI). The present study compared the effects of crushed ticagrelor vs. eptifibatide bolus + clopidogrel in troponin-negative ACS patients undergoing PCI.

DETAILED DESCRIPTION:
Platelet activation and accumulation causes the formation of blood clots that may cause heart attack. As a standard of care, the doctor can prescribe medications such as are ticagrelor, eptifibatide, clopidogrel, to prevent the formation of blood clots.

100 patients with unstable angina, both male and female, will be randomized to either Group A- Crushed Ticagrelor or Group B- Eptifibatide bolus +Clopidogrel administrated immediately before PCI. Platelet function testing, troponin, and ECG will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unstable angina/troponin negative ACS.

Exclusion Criteria:

1. need for oral anticoagulation therapy (Warfarin, Dabigatran, Rivaroxaban, Apixaban, Edoxaban)
2. increased risk of bradycardia, and the associated therapy with a strong cytochrome P-450 inhibitors (anti-retroviral agents, antifungal agents and some antibiotics eg. Indinavir, Nelfinavir, Lopinavir, Ritonavir, Itraconazole, Ketoconazole, Voriconazole, Clarithromycin, Telithormycin)
3. surgery<4 weeks
4. use of any thienopyridines (Clopidogrel, Prasugrel) 7 days prior to randomization
5. administration of GP IIb/IIIa inhibitors
6. bleeding diathesis or major bleeding episode within 2 weeks
7. thrombocytopenia (Platelet count < 100000)
8. incessant chest pain
9. hemodynamic instability (Mean arterial pressure < 65 mm Hg; need for vasopressor or inotropic agents; need for mechanical circulatory support for coronary intervention), NSTEMI as evidenced by elevation of troponin levels (Troponin > 0.034 ng/ml); renal failure with a serum creatinine >2.0 mg/dL
10. anemia with HCT<30%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massoud Leesar, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marian MJ, Abu Daya H, Chatterjee A, Al Solaiman F, Sasse MF, Fonbah WS, Workman RW, Johnson BE, Carlson SE, Brott BC, Prabhu SD, Leesar MA. Effects of Crushed Ticagrelor Versus Eptifibatide Bolus Plus Clopidogrel in Troponin-Negative Acute Coronary Syndrome Patients Undergoing Percutaneous Coronary Intervention: A Randomized Clinical Trial. J Am Heart Assoc. 2019 Dec 3;8(23):e012844. doi: 10.1161/JAHA.119.012844. Epub 2019 Nov 26. PMID 31766977

RESULTS

PARTICIPANT FLOW:
Groups:
- Eptifibatide Bolus+Clopidogrel: Eptifibatide bolus (180 mcg/kg x 2 boluses) + clopidogrel 600 mg and heparin low-dose (n=50 patients)
  Eptifibatide: After randomization, a blood sample will be obtained at baseline for platelet function test, the study drugs, clopidogrel and eptifibatide bolus will be administered. Patients will undergo PCI using drug-eluting stents or bare-metal stents. Blood samples will be obtained at 30 mins, 2, 4, and 24 h after PCI for platelet function tests.
  Clopidogrel
Period: Overall Study
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Started | 50 | 50
Completed | 50 | 48
Not Completed | 0 | 2
Not completed — blood samples hemolyzed | 0 | 2

BASELINE CHARACTERISTICS:
Population: 2 participants of the Eptifibatide Bolus+Clopidogrel arm were unable to be analyzed due to blood samples being hemolyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Number; unit: participants]
  >=19 years | 50 | 50 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 31 | 38 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in high-on Treatment Platelet Reactivity (HPR)
Description: We assessed platelet aggregation at baseline and during PCI by light transmission aggregomerty. The primary efficacy measure was HPR defined as platelet aggregation >59% at 2 h measured by the Chronlog aggregometer after stimulation with ADP 20 µM.
Time Frame: 5 times (at baseline, and at 0.5, 2, 4, and 24 hours after loading dose)
Population: as for baseline characteristics
Measure: Number; unit: count of participants
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 48
count of participants
  Baseline (n-50, n-48) | 37 | 33
  0.5 h (n-50, n-48) | 24 | 0
  2 h (n-50, n-48) | 6 | 0
  4 h (n-50, n-48) | 0 | 0
  24 h (n-50, n-48) | 2 | 5

2. Secondary Outcome: Number of Participants With a Periprocedural Myocardial Infarction and Injury (PMI)
Description: The rate of PMI will be compared in patients randomized to crushed ticagrelor vs. eptifibatide bolus +clopidogrel
Time Frame: At baseline and every 8 hours post- PCI
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
Participants | 24 | 14

3. Secondary Outcome: Platelet Aggregation Levels
Description: The rates of platelet aggregation with ADP and TRAP will be measured in patients randomized to crushed ticagrelor vs. eptifibatide bolus+clopidogrel
Time Frame: At baseline and at 0.5, 2, 4, and 24 hours after loading dose
Population: We did not have enough plasma sample to measure TRAP 10 at 4, 24 h.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 48
μmol/L
  Baseline (ADP 20) | 65 (14) | 62 (10)
  0.5 h (ADP 20) | 53 (12) | 1.3 (2)
  2 h (ADP 20) | 35 (11) | .34 (1)
  4 h (ADP 20) | 23 (9) | 3.5 (2)
  24 h (ADP 20) | 25 (10) | 38 (9)
  Baseline (ADP 5) | 56 (12) | 54 (13)
  0.5 h (ADP 5) | 44 (17) | 1.18 (4)
  2 h (ADP 5) | 24 (13) | .3 (.93)
  4 h (ADP 5) | 15 (9) | 1.6 (1.5)
  24 h (ADP 5) | 18 (14) | 27 (17)
  Baseline (TRAP 20) | 68 (14) | 67 (16)
  0.5 h (TRAP 20) | 60 (13) | 3.9 (3.6)
  2 h (TRAP 20) | 51 (8) | 6 (5)
  4 h (TRAP 20) | 48 (12) | 14 (10)
  24 h (TRAP 20) | 54 (11) | 51 (11)
  Baseline (TRAP 10) | 56 (18) | 54 (19)
  0.5 h (TRAP 10) | 48 (19) | 1.18 (1)
  2 h (TRAP 10) | 37 (17) | 1.57 (2)

4. Secondary Outcome: Change in Hemoglobin Levels (g/dL)
Description: Hemoglobin levels (g/dL) will be measured at baseline and on the next day after PCI.
Time Frame: At baseline and at 24 hours post-PCI
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
g/dL
  Baseline (hemoglobin, g/dL) | 13.52 (2) | 13.34 (1.62)
  Post-PCI (hemoglobin, g/dL) | 12.73 (1.81) | 12.71 (1.6)

5. Secondary Outcome: A Change in Hematocrit Levels
Description: Hematocrit levels (%) will be measured at baseline and on the next day after PCI.
Time Frame: At baseline and at 24 hours post-PCI
Measure: Mean (Standard Deviation); unit: hematocrit (%)
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
hematocrit (%)
  Baseline (hematocrit, %) | 40.11 (5.36) | 40.02 (4.49)
  Post-PCI (hematocrit, %) | 37.68 (4.85) | 37.5 (4.2)

6. Secondary Outcome: Heparin Dose, Unit/Kg
Description: For the heparin dose range for the two groups would have a minimum dose of 4693 and a maximum dose of 11141 units per kilogram.The higher the number is indicative that a higher dose of heparin is needed based on kilogram weight.
Time Frame: 24 hours after the PCI
Measure: Mean (Standard Deviation); unit: units per kilogram
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
units per kilogram | 8854 (2287) | 6021 (1328)

7. Secondary Outcome: Activated Clotting Time (ACT), Seconds
Description: The Level of the highest ACT during PCI will be compared between the groups
Time Frame: At the end of PCI
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
s | 332 (48) | 278 (47)

8. Secondary Outcome: Number of Patients With Minor Bleeding Complications
Description: We evaluated the number of patients with minor bleeding complications. Minor bleeding, based on Bleeding Academic Research Consortium (BARC), was defined as clinically overt (including imaging), resulting in hemoglobin drop of 3 to <5 g/dL.
Time Frame: At 24 hours post-PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

9. Secondary Outcome: Number of Patients With Minor Bleeding Complications
Description: as for outcome 8
Time Frame: At 1 year post-PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

10. Secondary Outcome: Number of Patients With Major Bleeding Complications
Description: We evaluated the number of patients with major bleeding complications. Major bleeding, based on Bleeding Academic Research Consortium (BARC), was defined as type 3a, bleeding + hemoglobin drop of 3 to <5 g/dL; type 3b, bleeding + hemoglobin drop ≥5 g/dL; and type C, intracranial hemorrhage.
Time Frame: At 24 hours post-PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

11. Secondary Outcome: Number of Patients With Major Bleeding Complications
Description: as for outcome 10
Time Frame: At 1 year post-PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

12. Secondary Outcome: Number of Patients With Negative Clinical Outcomes
Description: The rates of death, myocardial infarction, and revascularization at 1-year post-PCI.
Time Frame: At 1-year post-PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
Number analyzed (Participants) | 50 | 50
Participants
  Death | 2 | 0
  Myocardial infarction | 0 | 0
  Revascularization | 1 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks post-discharge
Arm/Group | Ticagrelor | Eptifibatide Bolus+Clopidogrel
All-Cause Mortality (participants affected / at risk) | 2/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=50) | Eptifibatide Bolus+Clopidogrel (N=50)
Target Lesion Revascularization (TLR) (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT02925923/Prot_SAP_000.pdf